CLINICAL TRIAL: NCT06287957
Title: Chitosan Brushes vs Air-Abrasive Devices on Peri-implant Mucositis Treatment: A Randomized Clinical
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Alper Gultekin, Dr., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IU-DHF-AG-01
Record Dates: First submitted 2024-02-24; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Peri-implant Mucositis; Peri-Implantitis; Bleeding on Probing; Periodontal Pocket
Keywords: peri-implant mucositis; Labrida Bioclean; Air-flow; Chitosan Brush; Peri-implantitis
MeSH Terms: conditions — Peri-Implantitis; Periodontal Pocket

STUDY DESIGN:
Intervention Model Description: There are going to be 4 treatment groups. Group 1: Mini Implant Platform treated with Labrida Bioclean Group 2: Regular Implant Platform treated with Labrida Bioclean Group 3: Mini Implant Platform treated with Air-Flow Device Group 4: Regular Implant Platform treated with Air-Flow Device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ML (Experimental): Patients with mini platform implants to be treated with Labrida Bioclean
  Interventions: Procedure: Labrida BioClean
- RL (Experimental): Patients with regular platform implants to be treated with Labrida Bioclean
  Interventions: Procedure: Labrida BioClean
- ME (Active Comparator): Patients with mini platform implants to be treated with Air-Flow Devices (EMS Handy 3.0 Perio Premium)
  Interventions: Procedure: EMS Handy 3.0 Perio Premium
- RE (Active Comparator): Patients with regular platform implants to be treated with Air-Flow Devices (EMS Handy 3.0 Perio Premium)
  Interventions: Procedure: EMS Handy 3.0 Perio Premium

INTERVENTIONS:
Procedure: Labrida BioClean — Debriding the tissue around the implant with Labrida Bioclean
  Arms: ML; RL
Procedure: EMS Handy 3.0 Perio Premium — Debriding the tissue around the implant with Air-Flow Device
  Arms: ME; RE

SUMMARY:
Bleeding on probing (0,1,2,3), plaque index (+,-) and pocket probing depth will be recorded for each visit. Before the procedure, the patient will be randomly assigned to one of four groups and records will be kept. In the frst visit of the patient, necessary actions will be taken according to the group to which the patient is assigned. The implant periphery of the patients assigned to the chitosan brush group will be debrided with a chitosan brush with circular movements. The implants of the patients assigned to the air abrasive device group will be cleaned in the same way with circular movements. The debrided area of both groups will be washed with sterile serum after the treatment. Patients will be called at the 2nd, 4th and 12th weeks and compared with the records kept.

DETAILED DESCRIPTION:
Patients with single implants and single cemented crowns with peri-implant mucositis on their posterior teeth (Premolars and molars) Regular peri-implant mucositis treatment with air-abrasive device and a new method with labrida bioclean brush for cleaning the infection.

Experimental procedures and follow-ups Bleeding on probing (0,1,2,3), plaque index (+,-) and pocket probing depth will be recorded for each visit. Before the procedure, the patient will be randomly assigned to one of four groups and records will be kept. In the frst visit of the patient, necessary actions will be taken according to the group to which the patient is assigned. The implant periphery of the patients assigned to the chitosan brush group will be debrided with a chitosan brush with circular movements. The implants of the patients assigned to the air abrasive device group will be cleaned in the same way with circular movements. The debrided area of both groups will be washed with sterile serum after the treatment. Patients will be called at the 2nd, 4th and 12th weeks and compared with the records kept.

The number of cases to be taken in total, 12 cases, was determined as 48. There will be 54-55 cases with 10% drop out share.

GPOWER PROTOCOL F tests - ANOVA: Repeated measures, between factors Analysis: A priori: Compute required sample size Input: Effect size f = 0.4982302 α err prob = 0.05 Power (1-β err prob) = 0.95 Number of groups = 4 Number of measurements = 4 Corr among rep measures = 0.5 Output: Noncentrality parameter λ = 19.0643199 Critical F = 2.8164658 Numerator df = 3.0000000 Denominator df = 44.0000000 Total sample size = 48 Actual power = 0.9529658 For the results; Data will be analyzed with IBM SPSS V23. Repeated measures analysis of variance will be used to analyze quantitative data. For multiple comparisons, the Bonferroni test will be used. Analysis results will be presented as mean and standard deviation for quantitative data, and frequency and percentage for categorical data. The signifcance level will be taken as p<0.05.

Peri-implant mucositis is the last reversible stage before peri-implantitis. Treatment of the disease at this stage is very important. When treated, bone loss around the implant will be prevented and implant survival will be prolonged.

ELIGIBILITY:
Inclusion Criteria:

* Presence of peri-implant mucositis around at least one implant,
* Being over 18 years old,
* Being psychologically suitable,
* The teeth adjacent to the relevant implant are natural teeth,
* Having at least 1 implant in the maxillary or mandibular posterior region (teeth 4, 5, 6 and 7) and a cemented prosthesis that is not connected to other implants or teeth as its superstructure,
* Probing depth longer than 3 mm and shorter than 5 mm,
* Evidence of bleeding is required on probing.

Exclusion Criteria:

* Pregnancy
* History of chemotherapy and/or radiotherapy received in the past or currently being received,
* Bone loss around the implant,
* Presence of an implant in the area adjacent to the relevant implant,
* Dentures combined with other implants or teeth,
* Screw-retained prostheses
* Uncontrolled diabetes

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Probing Depth | First visit, 2 weeks after the procedure, 4 weeks after the procedure, 8 weeks after the procedure
  Probing depth will be recorded for all around the implant on each visit of the patient. One of the inclusion criterias is 3 to 5 mm probing depth around the implant.

SECONDARY OUTCOMES:
Bleeding on Probing | First visit, 2 weeks after the procedure, 4 weeks after the procedure, 8 weeks after the procedure
  Bleeding on probing will be recorded on each visit of the patient (No bleeding 0, spot bleeding 1, Linear Bleeding 2, Bleeding all around 3).

OTHER OUTCOMES:
Plaque Index | First visit, 2 weeks after the procedure, 4 weeks after the procedure, 8 weeks after the procedure
  Plaque index will be recorded around the implant (+,-).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No